CLINICAL TRIAL: NCT00130806
Title: A Study to Assess the Efficacy and Tolerability of MK0478 (Muraglitazar, Also, BMS 298585) Coadministered With Insulin in Patients With Type 2 Diabetes
Brief Title: An Investigational Drug Co-Administered With Insulin in Patients With Type 2 Diabetes (0478-065)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0478-065; 2005_020
Record Dates: First submitted 2005-08-12; First posted 2005-08-16 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — muraglitazar

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0478 (muraglitazar)
Drug: Comparator: placebo

SUMMARY:
This is a study to evaluate the effectiveness and tolerability of an investigational drug in patients with type 2 diabetes (a specific type of diabetes) who are not currently treated with insulin.

DETAILED DESCRIPTION:
The duration of treatment is 30 weeks.

ELIGIBILITY:
Inclusion Criteria:

* People between the ages of 18 and 70 who have a specific type of diabetes called type 2 diabetes which is currently being treated only with oral medication(s). (Patients currently taking insulin would not be allowed to participate.)

Exclusion Criteria:

* People who have specific diseases (such as liver disease, gallbladder disease, pancreatitis, severe blood disorders or history of neoplastic diseases) which will be discussed by the study doctor and for which study participation would not be allowed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2005-09; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
The difference in daily dose requirements of insulin after 24 weeks

SECONDARY OUTCOMES:
(a) HbA1C; (b) FPG; (c) Percent of patients with HbA1C <7.0%; (d) TG, HDL-C, non-HDL-C and apolipoprotein B; (e) Free Fatty Acids (FFA); (f) the incidence of hypoglycemic events at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC